CLINICAL TRIAL: NCT03707067
Title: The Effects of Made-To-Measure Compression Garments on the Recovery of Performance and Markers of Muscle Damage and Inflammation in Elite Modern Pentathletes
Brief Title: Compression Garments for Recovery in Modern Pentathletes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St Mary's University College (Other)
Collaborators: Modern Pentathlon GB (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: SMU_SHAS_2018_02
Record Dates: First submitted 2018-06-07; First posted 2018-10-16 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-10

CONDITIONS: Muscle Damage
Keywords: exercise induced muscle damage; elite athlete; recovery

STUDY DESIGN:
Intervention Model Description: Crossover RCT
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomization carried out and compression garments allocated by a third party. All testing will be completed once athletes have removed their garments, without the knowledge of outcomes assessors or primary investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Custom fitted compression garments (Experimental): Made-to-measure compression garments providing high pressures (> 30 mmHg at the ankle and >20 mmHg at the thigh - equivalent to European class-2 stockings)
  Interventions: Device: Compression garments
- Sham recovery drink (Sham Comparator): Non-caloric beverage, labelled as a "recovery" drink to enhance athletic recovery. Aspartame/acesulfame-k based sweetener, providing 0.5 g carbohydrate and 2 Kcal per serving
  Interventions: Other: Sham recovery drink

INTERVENTIONS:
Device: Compression garments — Made-to-measure compression garments providing high pressures (> 30 mmHg at the ankle and >20 mmHg at the thigh - equivalent to European class-2 stockings)
  Arms: Custom fitted compression garments
Other: Sham recovery drink — Non-caloric beverage, labelled as a "recovery" drink proposed to enhance athletic recovery. Aspartame/acesulfame-k based sweetener, providing 0.5 g carbohydrate and 2 Kcal per serving
  Arms: Sham recovery drink

SUMMARY:
Aims To assess the efficacy of made to measure, high pressure compression garments (CG) for facilitating the recovery of strength, muscular power, and physiological markers of muscle damage following fencing, when compared a sham treatment

Rationale for study design

The results of a recent meta-analysis have informed the design of this study. The conclusions of the meta-analysis were that CG are most effective for the recovery of:

* Force and power performance following eccentric/plyometric exercise
* Maximal force production, at least 24 hours post-exercise (for example in strength and power athletes undertaking resistance training programmes)
* Additionally, the recovery of high-intensity cardiovascular performance may also be enhanced by the used of CG, when tested 24 hours following exercise which incurs metabolic stress Accordingly, the current study was designed to investigate the effects of CG of intense, competitive sparring following fencing sessions, held at the British Modern Pentathlon training base at the University of Bath.

DETAILED DESCRIPTION:
The efficacy of compression garments (CG) for recovery will be assessed in 10 elite modern pentathletes, using a crossover design. Athletes will complete each of two different recovery interventions immediately after each of 2 identical 3 hour fencing sessions, in a random order. Sessions will be separated by at least 2 weeks, standardising training in the lead-up to control for training-load and fatigue. A two-way (4 time-points x 2 conditions) crossover trial will be conducted to assess differences in performance tests following fencing ("sparring"), conducted before and after sparring, then 12 hours and 36 hours afterwards. In addition, 3200 m running performance will be assessed the afternoon before and at 12 hours and 36 hours after the fencing session.

All testing will be carried out at the British Modern Pentathlon base at the University of Bath. One month before testing, athletes will familiarised with strength testing using a strain-gauge (MIE Medical Research Ltd., Leeds, UK). Participants will be seated on a plyometric box, starting from a flexed position of 90 degrees, as measured with a goniometer, before taking the best of three attempts of maximal knee flexion. All other measures to be taken form part of the athletes' regular performance monitoring tests. Body composition will be assessed, including height and body-mass, as well as waist, hip thigh, calf, ankle and gluteal circumferences. All limb measurements will be taken from the right side, in accordance with guidelines set by the International Society of Anthropometry and Kinanthropometry (ISAK). Skinfold measurements will be taken according to the ISAK 8 site protocol by a level 1 anthropometrist. Athletes will be fitted for custom fitted (CF) CG (stockings), after taking real-time 3D images using the manufacturer's proprietary, digitised method (Isobar Compression Ltd., Manchester, UK).

In the afternoon before fencing begins (12 midday), 3200 m running performance will be timed using a stopwatch on a 400 m running track (8 laps). Fencing sparring will commence at 5 p.m. the same day, preceded immediately by the other performance measures and physiological tests. Following athletes' individual warm-ups, maximal leg strength will be assessed, as well as vertical jump performance (maximal force and maximum height from the best of 3 attempts) using a force plate (Kistler 3-Component Force-Link, New York, USA). Maximal grip strength will also be assessed (Takei Digital Hand-Grip Dynanometer 4001, Takei Scientific Instruments Co., Niigata-City, Japan). Soreness (200 mm visual analogue scale) and swelling at the mid-thigh skinfold site will also be recorded (spring loaded tape measure - Lafayette Instrument Co, Lafayette, Ind, USA). Muscle damage will be quantified with creatine kinase analysis (CK), and inflammation quantified with C-reactive protein (RX Daytona, Kearneysville, West Virginia, USA) from venous blood samples taken from the arm at baseline and at each time-point throughout recovery. Biomarkers of oxidative damage (the free oxygen radicals - FORT - test) and anti-oxidant defense (free oxygen radicals defense - FORD) will also be assessed. Testing will be conducted after warm-up before sparring, and then immediately after the cessation of the fencing session, after 12 hours and 36 hours recovery. However, 3200 m running performance will be assessed only in the afternoon before, then at 12 hours and 36 hours.

Athletes will complete each of two recovery conditions immediately after training and testing, being randomly assigned to a different condition over each session. Athletes will be allocated to one of the following 3 conditions:

* Custom fitted stockings applying over 30 mmHg and 20 mmHg at the calf and mid-thigh respectively (CF)
* A sham treatment (CON) The CON group will receive a sham "recovery" drink immediately after training (Robinsons no added sugar fruit juice), which contains 1 g carbohydrate and 0 g protein per serving. Pressures at the skin-garment interface will be measured for both garments using a pressure monitor at the medial calf and mid-thigh skinfold sites (as defined by the International Society for Anthropometry and Kinanthropometry), as well as 2 cm above the medial malleolus.

Between-treatment differences in the recovery of performance and physiological factors will be assessed over time using a 2 way (time by condition) mixed-measures analysis of variance (SPSS Statistics 22, IBM, New York, USA).

Equipment used and methods employed make use of validated measures of strength, power, muscle damage and compression pressures, cited in the protocol above.

ELIGIBILITY:
Inclusion Criteria:

* Athletes must be full-time athletes over the age of 18
* Training regularly for at least 3 months without extended disruption to training (> 2 weeks)

Exclusion Criteria:

* Presentation of injuries or chronic illnesses
* Inactivity or disruptions to training > 2 weeks (e.g. due to injury)
* The use of anti-inflammatory medications
* Over 40 years old (classification as a "Masters" athlete)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-11-30 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-02-28 (Estimated)

PRIMARY OUTCOMES:
Maximal isometric voluntary contraction strength for knee extension (change in Newtons compared to baseline) | 36 h. Second leg will be conducted after 1 week "washout" (10 days in total)
  Participants will be assessed for strength performance with maximal isometric voluntary contraction of the knee extensors (using a strain gauge) at the following time-points after fencing and compared to baseline: Immediately post, 12 hours post, 36 hours post-fencing (x 2 - crossover).
Lower body reactive strength (jump height/contact time in m/s) following a drop from a 0.6 m box onto a force plate (change in m/s compared to baseline) | 36 h. Second leg will be conducted after 1 week "washout" (10 days in total)
  Participants will be compared to baseline for reactive strength performance at the following time-points after fencing:Immediately post, 12 hours post, 36 hours post-fencing (x 2 - crossover).
  Jump height (m) and contact time (s) will be recorded following a drop from a 0.6 m box onto a force-plate.
3200 m run time trial performance (change in seconds compared to baseline) | 36 h. Second leg will be conducted after 1 week "washout" (10 days in total)
  Participants will be timed for 3200 m running performance at the following time-points after fencing and compared to baseline: Immediately post, 12 hours post, 36 hours post-fencing (x 2 - crossover).

SECONDARY OUTCOMES:
Perceived soreness, scored by drawing a vertical line on a 200 mm visual analogue scale from 0 mm (no soreness) to 200 mm (worst soreness imaginable). Change in mm will be compared to baseline. | 36 h. Second leg will be conducted after 1 week "washout" (10 days in total)
  Participants will be measured for muscular soreness at the following time-points after fencing and compared to baseline: Immediately post, 12 hours post, 36 hours post-fencing (x 2 - crossover). Perceived soreness will be scored by drawing a vertical line on a 200 mm visual analogue scale from 0 mm (no soreness) to 200 mm (worst soreness imaginable) and compared to baseline.
Circulating creatine kinase concentrations (CK - change in international units compared to baseline) | 36 h. Second leg will be conducted after 1 week "washout" (10 days in total)
  Participants will be measured for circulating creatine kinase concentrations (CK) at the following time-points after fencing and compared to baseline: Immediately post, 12 hours post, 36 hours post-fencing (x 2 - crossover). Change from baseline will be measured in international units (IU)
Mid-thigh girth (MTG) at the mid-thigh skinfold site as defined by International Society of Anthropometry and Kinanthropometry. Change will be measured in mm by comparing to baseline | 36 h. Second leg will be conducted after 1 week "washout" (10 days in total)
  Thigh circumference (mm) at the mid-thigh skinfold site (as defined by International Society of Anthropoemtry and Kinanthropometry) will be measured at the following time-points after fencing and compared to baseline: Immediately post, 12 hours post, 36 hours post-fencing (x 2 - crossover).
Free oxygen radicals defense (FORD) status (change in mmol/L Trolox equivalents compared to baseline) | 36 h. Second leg will be conducted after 1 week "washout" (10 days in total)
  Blood free oxygen radicals defense (FORD) will be measured from capillary samples taken from the earlobe at the following time-points after fencing and compared to baseline: Immediately post, 12 hours post, 36 hours post-fencing (x 2 - crossover).
Free oxygen radicals (FORT) status (change in mmol/L H2O2 equivalents compared to baseline) | 36 h. Second leg will be conducted after 1 week "washout" (10 days in total)
  Blood free oxygen radicals (FORT) will be measured from capillary samples taken from the earlobe at the following time-points after fencing and compared to baseline: Immediately post, 12 hours post, 36 hours post-fencing (x 2 - crossover).

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - University of Bath, Bath, Somerset
  - St Marys University, London

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol, Statistical Analysis Plan (SAP), Informed Consent Form (ICF) and Clinical Study Report (CSR) will all be available from February 2019
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Study Protocol, Statistical Analysis Plan (SAP), Informed Consent Form (ICF) and Clinical Study Report (CSR) will all be available from February 2019. Data will be stored for 10 years
Access Criteria: Must demonstrate planned research protocol and ethics application

REFERENCES:
- [Background] Brown F, Gissane C, Howatson G, van Someren K, Pedlar C, Hill J. Compression Garments and Recovery from Exercise: A Meta-Analysis. Sports Med. 2017 Nov;47(11):2245-2267. doi: 10.1007/s40279-017-0728-9. PMID 28434152
- [Background] Brophy-Williams N, Driller M, Halson S, Fell J, Shing C. Evaluating the Kikuhime pressure monitor for use with sports compression clothing. Sports Engineering. 2014;17(1):55-60